CLINICAL TRIAL: NCT07282314
Title: A Randomized Controlled Study on Autologous Platelet-rich Plasma Injection in Patients With Poor Ovarian Response
Brief Title: A RCT Study on Autologous PRP Injection in Patients With POR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Ma Caihong, Chief Physician, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00006761-M20250889
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Poor Ovarian Response; PRP Injection
Keywords: poor ovarian response; autologous platelet-rich plasma; Premature ovarian insufficiency
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP group (Experimental): Under ultrasound guidance, through vaginal puncture, PRP was injected subcutaneously into the ovarian cortex on both sides. There were 3 injection points on each side of the ovary, with 0.5ml injected at each point. The total injection volume for each side of the ovary was 1.5ml. The injection was carried out for 1 to 3 consecutive cycles.
  Interventions: Device: PRP injection
- Control Group (No Intervention): No intervention

INTERVENTIONS:
Device: PRP injection — Under ultrasound guidance, through vaginal puncture, PRP was injected subcutaneously into the ovarian cortex on both sides. There were 3 injection points on each side of the ovary, with 0.5ml injected at each point. The total injection volume for each side of the ovary was 1.5ml. The injection was carried out for 1 to 3 consecutive cycles.
  Arms: PRP group

SUMMARY:
Poor ovarian response (POR) is a pathological condition where the ovaries do not respond well to the stimulation of gonadotropins. It is mainly characterized by a low number of developing follicles, a high cancellation rate of the ovarian stimulation cycle, a small number of retrieved oocytes, and a low clinical pregnancy rate. Premature ovarian insufficiency (POI) is a special type of this condition and is one of the most difficult infertility diseases to treat. The incidence of POR and POI in reproductive-aged women in China is increasing year by year, making them key and challenging issues in reproductive medicine. Novel local ovarian cell therapy can improve the microenvironment for follicle development, promote the development and ovulation of "dormant" primordial follicles, and improve the quality of oocytes. This study intends to conduct a prospective randomized controlled trial to evaluate the safety and efficacy of autologous platelet-rich plasma (PRP) local injection therapy for improving ovarian reserve and IVF-ET outcomes in patients with POR and POI. This study is expected to improve the fertility of POR patients from the perspective of autologous cell therapy. The autologous PRP local injection technique does not involve ethical barriers, is easy to standardize the diagnosis and treatment process and operation system, and is suitable for clinical translation and promotion.

ELIGIBILITY:
Inclusion Criteria:

1. Women who have fertility requirements and are seeking IVF treatment at the Reproductive Medicine Center of Peking University Third Hospital
2. Age ≤ 45 years old, infertility duration ≥ 1 year
3. Meeting the diagnostic criteria for POI or the Poseidon diagnostic criteria for POR
4. Previous controlled ovarian stimulation resulted in no more than 3 oocytes retrieved and/or no transplantable embryos and/or previous embryo implantation failure ≥ 2 times
5. Uterus and bilateral adnexa are intact
6. BMI 18.5 - 29 kg/m²
7. Participants must have given informed consent for this study and voluntarily signed a written informed consent form.

Exclusion Criteria:

1. Congenital abnormalities of reproductive organs
2. Septicemia, platelet dysfunction syndrome and severe thrombocytopenia and other coagulation disorders or other hematological diseases
3. Suffering from autoimmune diseases or other endocrine disorders, with abnormal thyroid function and uncontrolled condition
4. Having a mass in the adnexal area with an unclear benign or malignant nature
5. Complicated with severe cardiovascular and cerebrovascular diseases, malignant tumors, hematological diseases and mental disorders, patients with impaired function of important organs
6. Those who have used systemic corticosteroids within the last 2 weeks, or used antiplatelet drugs such as aspirin within the last 48 hours
7. In the acute inflammatory stage
8. Those with a history of venous thrombosis or pulmonary embolism during the screening period

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 142 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of retrieved oocytes | 6 months
  The treatment is considered successful if the number of retrieved oocytes increases by ≥ 2 after the treatment. The effective rate of treatment = (number of effective treatment cycles) / (total number of cycles) × 100%

SECONDARY OUTCOMES:
Blood anti-Müllerian hormone (AMH) level | 6 months
  Treatment is considered successful if the AMH level rises continuously for two consecutive times. The effective rate of treatment = (number of effective cases) / (total number of cases) × 100%
Number of antral follicles | 6 months
  The treatment is considered successful if the number of antral follicles in both ovaries increases by ≥ 2 after treatment. The effective rate of treatment = (number of treated cases with effective results) / (total number of treated cases) × 100%
clinical pregnancy rate | 1 year